CLINICAL TRIAL: NCT00731692
Title: A Double-blind, Randomized, Multicenter, Placebo-controlled, Parallel-group Study Comparing the Efficacy and Safety of 0.5mg Fingolimod Administered Orally Once Daily Versus Placebo in Patients With Primary Progressive Multiple Sclerosis and An Open-label, Single-arm Extension Study to the Double-blind, Randomized, Multicenter, Placebo-controlled, Parallel-group Study Comparing the Efficacy and Safety of0.5 mg FTY720 Administered Orally Once Daily Versus Placebo in Patients With Primary Progressive Multiple Sclerosis
Brief Title: This Was an Open-label, Single-arm Extension Study (CFTY720D2306E1) to a Double-blind, Randomized Multicenter, Placebo-controlled, Parallel-group Core Study (CFTY720D2306) in PPMS.
Acronym: INFORMS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The extension study was terminated early after the results of the core study showed the study did not meet primary endpoint; confirmed disability progression
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CFTY720D2306; 2007-002627-32 (EudraCT Number); NCT01779934 (obsolete NCT alias)
Record Dates: First submitted 2008-08-07; First posted 2008-08-11 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Primary Progressive Multiple Sclerosis
Keywords: FTY720, primary progressive multiple sclerosis,PPMS
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- FTY720D 0.5 mg (Experimental): Cohort 2: The 0.5 mg group consists of patients who were directly randomized to fingolimod 0.5 mg (i.e. AFTER the amendment
  Interventions: Drug: FTY720
- Placebo (Placebo Comparator): Cohort 1 and 2: Patients randomized to placebo continued on placebo after re-randomization
  Interventions: Drug: Placebo
- FTY720D 1.25 mg switch to 0.5 mg (Experimental): Cohort 1: fingolimod 1.25 group consists of patients who were initially randomized to fingolimod 1.25 mg and switched to fingolimod 0.5 mg after amendment on Nov 2009
  Interventions: Drug: FTY720

INTERVENTIONS:
Drug: FTY720 — Fingolimod capsules at doses of 1.25 mg (prior to implementation of Amendment 5) and 0.5 mg (after Amendment 5) were administered orally once daily
  Arms: FTY720D 0.5 mg; FTY720D 1.25 mg switch to 0.5 mg
Drug: Placebo — Matching placebo capsules were administered orally once daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate whether FTY720 is effective in delaying MS disability progression compared to placebo in patients with PPMS. This was an open-label, single-arm extension study to a double-blind, randomized multicenter, placebo-controlled, parallel-group core study. The core study completed and eligible patients enrolled into the extension study at the next scheduled or unscheduled core study visit. All patients, regardless of their treatment in the core study, received fingolimod 0.5 mg in the extension study. The extension study was terminated early after the results of the core study became available showing that the study did not meet its primary endpoint which was defined as confirmed disability progression in this population

ELIGIBILITY:
Inclusion Criteria:

General

1. sign written informed consent prior to participating in the study
2. 25 through 65 years of age inclusive
3. females of childbearing potential must:

   * have a negative pregnancy test at Baseline (prior to randomization) and
   * use simultaneously two forms of effective contraception during the treatment and 3-months after discontinuation of study medication

Primary Progressive Multiple sclerosis.

1. diagnosis of primary progressive multiple sclerosis (according to the 2005 Revised McDonald criteria):
2. time since first reported symptoms between 2 and 10 years
3. evidence of clinical disability progression in the 2 years prior to Screening
4. disability status at Screening

   * EDSS score of 3.5-6.0 inclusive
   * pyramidal functional system score of 2 or more
   * 25'TWT less than 30 seconds

Extension study Inclusion criteria

* Patients initially randomized to fingolimod 1.25 mg or placebo as part of the first study cohort, were to have completed at least 3 years on study drug treatment at the time of extension study initiation.
* Patients initially randomized to fingolimod 0.5 mg or placebo as part of the second study cohort, were to have continued on study drug treatment until such time as the last ongoing patient enrolled in the study had reached 3 years in study

Exclusion Criteria:

PPMS specific:

* History of relapses/attacks
* Progressive neurological disorder other than PPMS
* Pure cerebellar syndrome or pure visual progressive syndrome or pure
* cognitive progressive syndrome
* Presence of spinal cord compression at screening MRI
* Relevant history of vitamin B12 deficit
* Evidence of syphilis or borreliosis at Screening

Cardiovascular conditions:

* Myocardial infarction within the past 6 months or current unstable ischemic heart disease
* History of angina pectoris due to coronary spasm or history of Raynaud's phenomenon
* Severe cardiac failure or cardiac arrest
* History of symptomatic bradycardia
* Resting pulse <55 bpm pre-dose
* History of sick sinus syndrome or sino-atrial heart block
* History or presence of second and third degree AV block or an increase QT interval (QTc>440 ms)
* Arrythmia requiring treatment with class III antiarrythmic drugs
* History of positive tilt test from workout of vasovagal syncope
* Hypertension, not controlled with medication

Pulmonary:

* Severe respiratory disease or pulmonary fibrosis
* TB
* Abnormal X-ray, suggestive of active pulmonary disease
* Abnormal PFT: <70% of predicted for FEV1 and FVC; <60% for DLCO
* Patients receiving chronic (daily) therapies for asthma

Hepatic:

* Known history of alcohol abuse, chronic liver or biliary disease
* Total or conjugated Brb >ULN, unless in context of Gilbert's syndrome
* AP >1.5xULN; ALT/AST >2xULN; GGT>3xULN

Other:

* History of chronic disease of the immune system other than MS
* Malignancy (other than successfully treated SCC or BCC)
* Diabetes Mellitus
* Macular Edema present at screening
* HIV, Hepatitis C or B, other active infection
* History of total lymphoid irradiation or bone marrow transplantation
* Serum creatinine >1.7 mg/dl
* WBC <3500 cells/mm3
* Lymphocyte count <800 cells/mm3
* History of substance abuse or any other factor that may interfere with subject ability to cooperate and comply with the study procedures
* Unable to undergo MRI scans
* Participation in any therapeutical clinical research study in the 6 months prior to randomization
* Pregnant or lactating women
* Drugs requiring wash-out period:

  3 months:
  * Systemic corticosteroids or ACTH
  * INF-beta

    6 months:
  * Immunosuppressive medication
  * Immunoglobulins
  * Monoclonal antibodies
* Drugs that exclude participation in the study:
* Cladribine
* Cyclophosphamide
* Mitoxantrone (except: patients who received a cumulative dose of no more than 60mg/m2 more than 5 years ago could enter the study)

Extension study Exclusion criteria

-Patients were not eligible for enrollment in the extension study if they had any of the following key exclusion criteria at the extension study Baseline visit: active chronic immune system disease other than MS (or stable disease treated with immune therapy); known immunodeficiency syndrome; active infection; uncontrolled diabetes mellitus; macularedema; treatment with Class Ia or III antiarrhythmic drugs; any of the specified cardiac, pulmonary, or hepatic conditions; or any medically unstable condition

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 970 (Actual)
Dates: Start 2008-07-28 (Actual); Primary Completion 2015-06-22 (Actual); Study Completion 2015-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (143):
- United States (32):
  - Novartis Investigative Site, Newport Beach, California
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, Aurora, Colorado
  - Novartis Investigative Site, Pompano Beach, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Kansas City, Kansas
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Brookline, Massachusetts
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Teaneck, New Jersey
  - Novartis Investigative Site, Buffalo, New York
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Rochester, New York
  - Novartis Investigative Site, Stony Brook, New York
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Durham, North Carolina
  - Novartis Investigative Site, Cleveland, Ohio
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, Knoxville, Tennessee
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Burlington, Vermont
  - Novartis Investigative Site, Charlottesville, Virginia
  - Novartis Investigative Site, Seattle, Washington
  - Novartis Investigative Site, Madison, Wisconsin
- Australia (6):
  - Novartis Investigative Site, Camperdown, New South Wales
  - Novartis Investigative Site, Liverpool, New South Wales
  - Novartis Investigative Site, Hobart, Tasmania
  - Novartis Investigative Site, Box Hill, Victoria
  - Novartis Investigative Site, Heidelberg, Victoria
  - Novartis Investigative Site, Parkville, Victoria
- Belgium (6):
  - Novartis Investigative Site, Charleroi
  - Novartis Investigative Site, Edegem
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
  - Novartis Investigative Site, Melsbroek
  - Novartis Investigative Site, Sint-Truiden
- Canada (11):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Burnaby, British Columbia
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Gatineau, Quebec
  - Novartis Investigative Site, Greenfield Park, Quebec
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Regina, Saskatchewan
- Czechia (7):
  - Novartis Investigative Site, Brno, Czech Republic
  - Novartis Investigative Site, Rychnov nad Kněžnou, Czech Republic
  - Novartis Investigative Site, Olomouc, CZE
  - Novartis Investigative Site, Ostrava-Poruba
  - Novartis Investigative Site, Pilsen
  - Novartis Investigative Site, Prague
  - Novartis Investigative Site, Teplice
- Denmark (2):
  - Novartis Investigative Site, Aarhus
  - Novartis Investigative Site, Sønderborg
- Finland (3):
  - Novartis Investigative Site, Helsinki
  - Novartis Investigative Site, Tampere
  - Novartis Investigative Site, Turku
- France (8):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Strasbourg
- Germany (15):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Hennigsdorf
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Teupitz
  - Novartis Investigative Site, Trier
  - Novartis Investigative Site, Würzburg
- Hungary (5):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Győr
  - Novartis Investigative Site, Miskolc
  - Novartis Investigative Site, Veszprém
- Italy (11):
  - Novartis Investigative Site, Bari, BA
  - Novartis Investigative Site, Montichiari, BS
  - Novartis Investigative Site, Chieti, CH
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Cefalù, PA
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Orbassano, TO
  - Novartis Investigative Site, Gallarate, VA
- Netherlands (6):
  - Novartis Investigative Site, Breda, CK
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Eindhoven
  - Novartis Investigative Site, Nieuwegein
  - Novartis Investigative Site, Nijmegen
  - Novartis Investigative Site, Sittard-Geleen
- Poland (3):
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Lublin
  - Novartis Investigative Site, Warsaw
- Spain (10):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Bilbao, Basque Country
  - Novartis Investigative Site, Badalona, Catalonia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Girona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, Lleida, Catalonia
  - Novartis Investigative Site, Majadahonda, Madrid
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Madrid
- Sweden (2):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Stockholm
- Switzerland (5):
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Lausanne
  - Novartis Investigative Site, Lugano
  - Novartis Investigative Site, Zurich
- Turkey (Türkiye) (5):
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Atakum / Samsun
  - Novartis Investigative Site, Balcova / Izmir
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Yenisehir / Izmir
- United Kingdom (6):
  - Novartis Investigative Site, Salford, Manchester
  - Novartis Investigative Site, Sheffield, South Yorkshire
  - Novartis Investigative Site, Bristol
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Newcastle upon Tyne
  - Novartis Investigative Site, Norwich

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Calvi A, Mendelsohn Z, Hamed W, Chard D, Tur C, Stutters J, MacManus D, Kanber B, Wheeler-Kingshott CAMG, Barkhof F, Prados F. Treatment reduces the incidence of newly appearing multiple sclerosis lesions evolving into chronic active, slowly expanding lesions: A retrospective analysis. Eur J Neurol. 2024 Jan;31(1):e16092. doi: 10.1111/ene.16092. Epub 2023 Oct 12. PMID 37823722
- [Derived] Leppert D, Kropshofer H, Haring DA, Dahlke F, Patil A, Meinert R, Tomic D, Kappos L, Kuhle J. Blood Neurofilament Light in Progressive Multiple Sclerosis: Post Hoc Analysis of 2 Randomized Controlled Trials. Neurology. 2022 May 24;98(21):e2120-e2131. doi: 10.1212/WNL.0000000000200258. Epub 2022 Apr 4. PMID 35379762
- [Derived] Koch MW, Mostert J, Repovic P, Bowen JD, Strijbis E, Uitdehaag B, Cutter G. Smoking, obesity, and disability worsening in PPMS: an analysis of the INFORMS original trial dataset. J Neurol. 2022 Mar;269(3):1663-1669. doi: 10.1007/s00415-021-10750-z. Epub 2021 Aug 15. PMID 34392376
- [Derived] Koch MW, Mostert J, Zhang Y, Wolinsky JS, Lublin FD, Strijbis E, Cutter G. Association of Age With Contrast-Enhancing Lesions Across the Multiple Sclerosis Disease Spectrum. Neurology. 2021 Sep 28;97(13):e1334-e1342. doi: 10.1212/WNL.0000000000012603. Epub 2021 Aug 10. PMID 34376508
- [Derived] Miller DH, Lublin FD, Sormani MP, Kappos L, Yaldizli O, Freedman MS, Cree BAC, Weiner HL, Lubetzki C, Hartung HP, Montalban X, Uitdehaag BMJ, MacManus DG, Yousry TA, Gandini Wheeler-Kingshott CAM, Li B, Putzki N, Merschhemke M, Haring DA, Wolinsky JS. Brain atrophy and disability worsening in primary progressive multiple sclerosis: insights from the INFORMS study. Ann Clin Transl Neurol. 2018 Jan 30;5(3):346-356. doi: 10.1002/acn3.534. eCollection 2018 Mar. PMID 29560379
- [Derived] Lublin F, Miller DH, Freedman MS, Cree BAC, Wolinsky JS, Weiner H, Lubetzki C, Hartung HP, Montalban X, Uitdehaag BMJ, Merschhemke M, Li B, Putzki N, Liu FC, Haring DA, Kappos L; INFORMS study investigators. Oral fingolimod in primary progressive multiple sclerosis (INFORMS): a phase 3, randomised, double-blind, placebo-controlled trial. Lancet. 2016 Mar 12;387(10023):1075-1084. doi: 10.1016/S0140-6736(15)01314-8. Epub 2016 Jan 28. PMID 26827074
- [Derived] Hartung HP, Aktas O. Bleak prospects for primary progressive multiple sclerosis therapy: downs and downs, but a glimmer of hope. Ann Neurol. 2009 Oct;66(4):429-32. doi: 10.1002/ana.21880. No abstract available. PMID 19847907

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were randomized equally to receive either fingolimod or placebo. Patients initially randomized to fingolimod 1.25 mg/day or matching placebo groups switched in a blinded manner to fingolimod 0.5 mg/day or continued on placebo after amendment in Nov. 2009. Patients were randomized to receive either fingolimod 0.5 mg/day or placebo..
Pre-assignment Details: Prior to protocol amendment 147 patients received 1.25mg of FTY720; post protocol amendment 5 not all 147 patients switched to 0.5mg FTY720, only 121 switched and their data is presented under the 0.5mg dose.
Groups:
- FTY720 1.25 mg to 0.5 mg: Cohort 1: fingolimod 1.25 group consists of patients who were initially randomized to fingolimod 1.25 mg and switched to fingolimod 0.5 mg after amendment
- FTY720 0.5 mg to 0.5 mg: Cohort 2: The 0.5 mg group consists of patients who were directly randomized to fingolimod 0.5 mg (i.e. AFTER the amendment)
- Placebo to -FTY 0.5 mg: Cohort 1 and 2: Patients who started on placebo continued on placebo after re-randomization
Period: Core Study (36 Months)
Arm/Group | FTY720 1.25 mg to 0.5 mg | FTY720 0.5 mg to 0.5 mg | Placebo to -FTY 0.5 mg
Started | 147 | 336 | 487
Safety Set (SAF) | 0 | 336 | 487
Full Analysis Set (FAS) | 0 | 336 | 487
Pharmacokinetic Analysis Set | 102 | 249 | 0
Post Protocol Amendment 5 Switch | 0 | 121 (post protocol amendment 121 patients switch to 0.5 mg dose from 125mg dose) | 0
Completed | 79 | 220 | 317
Not Completed | 68 | 116 | 170
Not completed — Lack of Efficacy | 11 | 23 | 64
Not completed — Physician Decision | 1 | 0 | 2
Not completed — Death | 2 | 1 | 2
Not completed — Lost to Follow-up | 1 | 3 | 3
Not completed — Administrative | 2 | 2 | 6
Not completed — Abnormal Test Procedure Result | 4 | 3 | 5
Not completed — Protocol Violation | 4 | 5 | 8
Not completed — Abnormal Lab values | 6 | 19 | 5
Not completed — Adverse Event | 25 | 28 | 29
Not completed — Withdrawal by Subject | 12 | 32 | 46
Period: Extension Phase
Arm/Group | FTY720 1.25 mg to 0.5 mg | FTY720 0.5 mg to 0.5 mg | Placebo to -FTY 0.5 mg
Started | 74 | 196 | 301
Completed | 0 | 0 | 0
Not Completed | 74 | 196 | 301
Not completed — Admin Problems: Terminated # patients | 69 | 189 | 277
Not completed — Abnormal test procedure | 0 | 0 | 1
Not completed — Abnormal lab values | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 4
Not completed — Withdrawal by Subject | 4 | 5 | 3
Not completed — Adverse Event | 1 | 1 | 15

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Cohort 1 and 2: Patients who started on placebo continued on placebo after re-randomization
- Total: Total of all reporting groups
Arm/Group | FTY720 1.25 mg to 0.5 mg | FTY720 0.5 mg to 0.5 mg | Placebo | Total
Number analyzed (Participants) | 147 | 336 | 487 | 970
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (8.47) | 48.5 (8.59) | 48.5 (8.31) | 48.5 (8.42)
Age, Customized [Number; unit: Particpants]
  <=30 | 3 | 6 | 4 | 13
  31 to 40 | 22 | 60 | 90 | 172
  41 to 50 | 68 | 127 | 194 | 389
  >50 | 54 | 143 | 199 | 396
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 163 | 235 | 469
  Male | 76 | 173 | 252 | 501

OUTCOME MEASURES:

1. Primary Outcome: Kaplan-Meier Estimate of the Risk of 3-month Confirmed Disability Progression Based on Composite Endpoint
Description: 3-month sustained increase from Baseline in EDSS (at least 1 point increase from Baseline for patients with a Baseline value of 5 or less or at least 0.5 point increase from Baseline for patients with a Baseline value of 5.5 or more) or 3-month sustained increase of at least 20% from BL in the time taken to complete the timed 25-foot walk test (25' TWT); or 3-month sustained increase of at least 20% from BL in the time taken to complete the 9-HPT. The 25' TWT is a quantitative measure of lower extremity function. The EDSS is a scale assessing neurologic impairment, including a series of scores in each of 8 functional systems: Visual, Brain Stem, Pyramidal, Cerebellar, Sensory, Bowel and Bladder, Cerebral and Other functions. The score ranges from 0 (normal) to 10 (death due to MS)). The 9-hole peg test (9-HPT) is a quantitative measure of upper extremity (arm and hand) function.
Time Frame: up to 36 months after the last patient was randomized
Population: Full analysis set (FAS) - The main efficacy analyses were performed using the FAS, in patients who were initially randomized to either FTY 0.5mg or to Placebo.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | FTY720 0.5 mg to 0.5 mg | Placebo
Number analyzed (Participants) | 336 | 487
Percentage of Participants | 77.2 [71.87 to 82.51] | 80.3 [73.31 to 87.25]
Statistical Analysis 1: Comparison: FTY720 0.5 mg to 0.5 mg vs Placebo; Test type: Superiority or Other; p = 0.544, Regression, Cox; Cox Proportional Hazard = 0.95, 95% CI 2-sided [0.80 to 1.12]

2. Secondary Outcome: Kaplan-Meier Estimate of the Risk of 3- Month Confirmed Disability Progression Based on Expanded Disability Status Scale (EDSS)
Description: The Expanded Disability Status Scale (EDSS) is a scale for assessing neurologic impairment in MS (Kurtzke 1983) and includes a series of scores in each of 8 functional systems and the EDSS steps (ranging from 0 (normal) to 10 (death due to MS)). The functional systems are Visual, Brain Stem, Pyramidal, Cerebellar, Sensory, Bowel and Bladder, Cerebral and Other functions. Fatigue is not included in the Cerebral score of the EDSS. The score ranges from 0 (normal) to 10 (death due to MS)
Time Frame: up to 36 months after the last patient was randomized
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | FTY720 0.5 mg to 0.5 mg | Placebo
Number analyzed (Participants) | 336 | 487
Percentage of Participants | 54.3 [47.16 to 61.45] | 58.7 [53.30 to 64.18]

3. Secondary Outcome: Percent Change From Baseline in Brain Volume at Month 36
Description: The percent change from Baseline in brain volume was analyzed using a random coefficients model. The model included: 1) fixed effects: treatment and region and 2) continuous covariates: time, number of Gd enhancing lesions at Baseline, Baseline T2 volume, and normalized brain volume at Baseline. Time as a continuous covariate allowed for the estimation of different slopes and intercepts among treatment groups.
Time Frame: Baseline to month 36
Population: Full analysis set (FAS) - The main efficacy analyses were performed using the FAS, in patients who were initially randomized to either FTY 0.5mg or to Placebo. N= Total number of patients included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | FTY720 0.5 mg to 0.5 mg | Placebo
Number analyzed (Participants) | 293 | 421
Percent Change | -1.49 [-1.64 to -1.35] | -1.53 [-1.65 to -1.41]

4. Secondary Outcome: Kaplan Meier Estimate -Percentage of Participants With 3- Month Confirmed Disability Progression Based on 9-HPT.
Description: The 9-HPT is a quantitative measure of upper extremity (arm and hand) function designed and validated for evaluation of MS patients. N= Total number of patients included in the analysis
Time Frame: up to 36 months after the last patient was randomized
Population: as for outcome 1
Measure: Number; unit: Percentge of Participants
Arm/Group | FTY720 0.5 mg to 0.5 mg | Placebo
Number analyzed (Participants) | 147 | 133
Percentge of Participants | 25.0 | 24.9

5. Secondary Outcome: Kaplan Meier Estimate -Percentage of Participants With 3- Month Confirmed Disability Progression Based on 25' TWT.
Description: The 25' TWT is a quantitative measure of lower extremity function designed and validated for evaluation of MS patients. N= Total number of patients included in the analysis
Time Frame: up to 36 months after the last patient was randomized
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | FTY720 0.5 mg to 0.5 mg | Placebo
Number analyzed (Participants) | 147 | 133
Percentage of Participants | 54.8 | 56.7

6. Secondary Outcome: Number of New/Enlarging T2 Lesions Per Year Measured From Baseline to Month 36
Description: Inflammatory disease, as measured by number of new or newly-enlarging T2 lesions, was assessed by Magnetic resonance Imaging (MRI) scanning of the brain and full spinal cord. N= Total number of patients included in the analysis
Time Frame: Baseline to 36 months
Population: Full analysis set (FAS) -The main efficacy analyses were performed using the FAS, in patients who were initially randomized to either FTY 0.5mg or to Placebo.
Measure: Least Squares Mean (95% Confidence Interval); unit: T2 Lesions per year
Arm/Group | FTY720 0.5 mg to 0.5 mg | Placebo
Number analyzed (Participants) | 298 | 421
T2 Lesions per year | 0.13 [0.10 to 0.18] | 0.50 [0.40 to 0.61]

7. Secondary Outcome: Number of Gd-enhancing Lesions at Month 36
Description: Inflammatory disease, as measured by number of T1 Gd-enhancing lesions, was assessed by MRI scanning of the brain and full spinal cord. N= Total number of patients included in the analysis
Time Frame: Baseline to 36 months
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Gd-enhanced lesions per patient per scan
Arm/Group | FTY720 0.5 mg to 0.5 mg | Placebo
Number analyzed (Participants) | 223 | 320
Gd-enhanced lesions per patient per scan | 0.05 [0.02 to 0.09] | 0.21 [0.15 to 0.30]

8. Secondary Outcome: Percent Change in Total T2 Lesion Volume From Baseline to Month 36
Description: Inflammatory disease as measured by percent change in total T2 lesion volume (mm3) was assessed by MRI. N= Total number of patients included in the analysis
Time Frame: Baseline to month 36
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | FTY720 0.5 mg to 0.5 mg | Placebo
Number analyzed (Participants) | 224 | 326
Percent Change | -9.2 (30.55) | 8.9 (44.13)

9. Secondary Outcome: Change From Baseline in the Patient Reported Indices in Multiple Sclerosis (PRIMUS-QoL Score)
Description: The quality of life scale contains 22 items. Each item will be given a score of 1 or 0. A score of 1 (or 0) indicates the presence (or absence) of the symptom or adverse quality of life. All 22 item scores will be summed to obtain a total score ranging from 0 (good) to 22 (poor), which is the PRIMUS QoL scale score
Time Frame: Baseline, 36 months
Population: Full analysis set (FAS) - The main efficacy analyses were performed using the FAS, in patients who were initially randomized to either FTY 0.5mg or to Placebo. Only subjects with a value at both baseline and at month 36 are included.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | FTY720 1.25 mg to 0.5 mg | FTY720 0.5 mg to 0.5 mg | Placebo
Number analyzed (Participants) | 66 | 150 | 230
Score on a scale | 0.2424 (4.18444) | 0.5921 (4.77704) | 0.9597 (4.38578)

10. Secondary Outcome: Change From Baseline in PRIMUS-Activities
Description: The activities subscale of PRIMUS contains 15 items and each item is given a score of 0 (able to do on own without difficulties), 1 (able to do on own with difficulties), or 2 (unable to do on own). All 15 items were summed to obtain a total score ranging from 0 (good) to 30 (poor).
Time Frame: Baseline, 36 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | FTY720 1.25 mg to 0.5 mg | FTY720 0.5 mg to 0.5 mg | Placebo
Number analyzed (Participants) | 68 | 153 | 237
Score on a scale | 3.5504 (7.05241) | 2.6324 (6.22256) | 2.8830 (6.76499)

11. Secondary Outcome: Change From Baseline in Unidimensional Fatigue Impact (U-FIS) Score
Description: Unidimensional Fatigue Impact Scale (U-FIS), contains 22 patient-reported items that assess the impact of fatigue on cognitive, physical, and psychosocial functioning. Responses formed a single unidimensional scale measuring fatigue impact. The U-FIS was calculated and analyzed according to the U-FIS scoring manual. The U-FIS scale contains 22 items with 5 possible outcomes for each item. Two response categories (about half the time and a lot of the time) were combined into 1 category to obtain 4 possible outcomes: 0 (never), 1 (a little of the time), 2 (about half the time/a lot of the time), and 3 (all the time). The 22 condensed item scores were summed to obtain a total score ranging from 0 (no fatigue) to 66 (severe fatigue impact).
Time Frame: Baseline, 36 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | FTY720 1.25 mg to 0.5 mg | FTY720 0.5 mg to 0.5 mg | Placebo
Number analyzed (Participants) | 70 | 154 | 241
Score on a scale | 1.3197 (12.44042) | 2.8451 (14.04769) | 3.1394 (12.20929)

12. Secondary Outcome: Change From Baseline in European Quality of Life - 5 Dimensions (EQ-5D Score)
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state (confined to bed). Scoring formula developed by EuroQoL Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state.
Time Frame: Baseline, 36 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | FTY720 1.25 mg to 0.5 mg | FTY720 0.5 mg to 0.5 mg | Placebo
Number analyzed (Participants) | 99 | 213 | 320
Score on a scale | -0.0332 (0.19420) | -0.0475 (0.26099) | -0.0539 (0.22383)

13. Secondary Outcome: Change From Baseline in Multiple Sclerosis Walking Scale (MSWS-12 Score)
Description: The Multiple Sclerosis Walking Scaleis a patient reported measure of walking quality (Hobart et al 2003), consisting of 12 items asking patients to rate the impact of MS upon their walking ability. Responses were captured on a 3-point scale ranging from 1 (Not at all) to 3 (A lot) for items 1 to 3 and on a 5-point scale ranging from 1 (not limited) to 5 (extremely) for items 4 to 12. All 12 item scores were summed to obtain a total score ranging from 12 (good) to 54 (poor) which is the MSWS-12 scale score. The total score was transformed to a 0 to 100 scale score. The MSWS-12 scale score will be transformed to a 0-100 scale score before any summaries or statistical analyses are performed. The transformed score is obtained by subtracting 12 and divided by 42 and multiplying by 100 (i.e., transformed scale score = (raw scale score- 12)/42*100).
Time Frame: Baseline, 36 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | FTY720 1.25 mg to 0.5 mg | FTY720 0.5 mg to 0.5 mg | Placebo
Number analyzed (Participants) | 75 | 182 | 261
Score on a scale | 6.4444 (23.81568) | 5.5616 (24.59030) | 9.5899 (23.98316)

14. Secondary Outcome: Blood Concentrations of Fingolimod and Fingolimod-phosphate
Description: Concentrations of fingolimod and fingolimod-phosphate in whole blood were determined by validated liquid chromatography methods with tandem mass spectrometry. The lower limits of quantification were 0.08 ng/ml for fingolimod and 0.1 ng/ml for fingolimod-phosphate.
  Venous blood samples were collected for the analysis.
Time Frame: Month 3 up to 36 months
Population: Full analysis set (FAS) -The main efficacy analyses were performed using the FAS, in patients who were initially randomized to either FTY 0.5mg or to Placebo. (N). Only participants (n) who provided one or more evaluable blood concentration were included in the pharmacokinetic analysis population. Analysis include 147 patients (cohort 1)
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- FTY720 1.25mg to 0.5 mg: fingolimod 1.25mg/0.5 mg group consists of patients who were initially randomized to fingolimod 1.25 mg and switched to fingolimod 0.5 mg
Arm/Group | FTY720 1.25 mg to 0.5 mg | FTY720 1.25mg to 0.5 mg | FTY720 0.5 mg to 0.5 mg
Number analyzed (Participants) | 102 | 102 | 249
ng/ml
  Month 3 Fingolimod (n=64, 179) | 6.04 (3.11) | NA (NA) — No evaluable blood concentration available | 2.58 (1.34)
  Month 12 Fingolimod (n=23, 161) | 6.24 (2.21) | 2.87 (1.70) | 2.55 (1.37)
  Month 18 Fingolimod (n=71,155) | NA (NA) — Patients switched to 0.5mg. No evaluable blood concentration available | 2.44 (1.15) | 2.59 (1.44)
  Month 24 Fingolimod (n=67, 160) | NA (NA) — Patients switched to 0.5mg. No evaluable blood concentration available | 2.41 (1.30) | 2.64 (1.50)
  Month 30 Fingolimod (n=62, 158) | NA (NA) — Patients switched to 0.5mg. No evaluable blood concentration available | 2.52 (1.28) | 2.60 (1.33)
  Month 36 Fingolimod (n=55, 118) | NA (NA) — Patients switched to 0.5mg. No evaluable blood concentration available | 2.44 (1.08) | 2.63 (1.38)
  End of treatment Fingolimod (n=32, 115) | NA (NA) — Patients switched to 0.5mg. No evaluable blood concentration available | 2.02 (1.10) | 2.57 (1.51)
  Month 3 Fingolimod-Phosphate (n=64, 179) | 3.20 (1.73) | NA (NA) — No evaluable blood concentration available | 1.40 (0.747)
  Month 12 Fingolimod-Phosphate (n=23, 161) | 3.21 (1.16) | 1.54 (0.871) | 1.43 (0.805)
  Month 18 Fingolimod-Phosphate (n=71,155) | NA (NA) — Patients switched to 0.5mg. No evaluable blood concentration available | 1.34 (0.630) | 1.41 (0.758)
  Month 24 Fingolimod-Phosphate (n=67, 160) | NA (NA) — Patients switched to 0.5mg. No evaluable blood concentration available | 1.35 (0.765) | 1.44 (0.790)
  Month 30 Fingolimod-Phosphate (n=62, 158) | NA (NA) — Patients switched to 0.5mg. No evaluable blood concentration available | 1.32 (0.676) | 1.48 (0.759)
  Month 36 Fingolimod-Phosphate (n=55, 118) | NA (NA) — Patients switched to 0.5mg. No evaluable blood concentration available | 1.32 (0.591) | 1.51 (0.765)
  End of treatment Fingolimod-Phosphate (n=32, 115 | NA (NA) — Patients switched to 0.5mg. No evaluable blood concentration available | 1.19 (0.618) | 1.50 (0.900)

15. Secondary Outcome: Change in MSFC Z-score and Subscale Scores From Baseline to Month 36
Description: The Multiple Sclerosis Functional Composite (MSFC) is a multidimensional clinical outcome measure that includes quantitative tests of leg function/ambulation (Timed 25-Foot Walk), arm function (9-Hole Peg Test), and cognitive function (Paced Auditory Serial Addition Test). The overall MSFC z-score as an average of the three standardized scores derived using baseline data pooled over each treatment arm as reference population. Higher scores reflect better neurological function and a positive change from Baseline indicates improvement.
Time Frame: Baseline to Month 36
Population: Full analysis set (FAS) - The main efficacy analyses were performed using the FAS
Measure: Mean (Standard Deviation); unit: Z-scores
Groups:
- FTY720 0.5 mg: Cohort 2: The 0.5 mg group consists of patients who were directly randomized to fingolimod 0.5 mg (i.e. AFTER the amendment)
Arm/Group | FTY720 0.5 mg | Placebo
Number analyzed (Participants) | 193 | 279
Z-scores | -0.189 (0.6980) | -0.212 (0.8468)

ADVERSE EVENTS:
Groups:
- Core: FTY720 1.25 mg: Patients who received FTY720 1.25 mg during core
- Core: FTY720 0.5 mg: Patients who received FTY720 0.5 mg during core
- Core: Placebo: Patients who received Placebo during core
- Extension: FTY1.25-0.5: Patients who received FTY20 1.25 mg in core and received 0.5 mg of FTY during Extension
- Extension: FTY0.5-0.5: Patients who received FTY20 0.5 mg in core and received 0.5 mg of FTY during Extension
- Extension: Placebo-FTY0.5: Patients who received Placebo in core and received 0.5 mg of FTY during Extension
Arm/Group | Core: FTY720 1.25 mg | Core: FTY720 0.5 mg | Core: Placebo | Extension: FTY1.25-0.5 | Extension: FTY0.5-0.5 | Extension: Placebo-FTY0.5
Serious Adverse Events (participants affected / at risk) | 38/147 | 84/336 | 117/487 | 7/74 | 10/196 | 37/301
Other Adverse Events (participants affected / at risk) | 132/147 | 278/336 | 406/487 | 43/74 | 70/196 | 138/301
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Core: FTY720 1.25 mg (N=147) | Core: FTY720 0.5 mg (N=336) | Core: Placebo (N=487) | Extension: FTY1.25-0.5 (N=74) | Extension: FTY0.5-0.5 (N=196) | Extension: Placebo-FTY0.5 (N=301)
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1
Atrioventricular block (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 2 | 2 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tachycardia paroxysmal (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0
Amblyopia strabismic (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Angle closure glaucoma (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cataract cortical (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Chorioretinopathy (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cystoid macular oedema (Eye disorders) | 0 | 1 | 1 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Intraocular haematoma (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Macular oedema (Eye disorders) | 1 | 4 | 4 | 0 | 0 | 0
Myopia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Optic atrophy (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 1 | 1 | 0 | 0 | 0
Retinal tear (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Anal polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Obstruction gastric (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 1 | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Device dislocation (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Device occlusion (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Drug ineffective (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 1 | 0 | 0 | 1
Gait disturbance (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
General physical health deterioration (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 3 | 0 | 0 | 0
Cholelithiasis obstructive (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 2 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Blister infected (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Bursitis infective (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 0
Dengue fever (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0
Enterocolitis bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Epididymitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 2 | 1 | 0 | 0 | 0
H1N1 influenza (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 2 | 1 | 0 | 0 | 0
Herpes zoster infection neurological (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Herpes zoster meningomyelitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Incision site infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 3 | 0 | 0 | 0 | 1
Meningitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Myelitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Ophthalmic herpes simplex (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 2 | 4 | 2 | 1 | 0 | 1
Pulmonary sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 3 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Serratia sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Systemic mycosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Tracheobronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 8 | 12 | 1 | 0 | 4
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 2 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 1 | 3 | 0 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1 | 3 | 0 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Fracture displacement (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1
Traumatic renal injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Foetal heart rate abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
International normalised ratio decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Troponin increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 2
Bone swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 11 | 9 | 1 | 2 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0 | 1 | 0 | 0
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Medullary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Metastases to kidney (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0
Osteoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0 | 0
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 6 | 1 | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Arachnoiditis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Central nervous system lesion (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0
Cerebrovascular disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Monoparesis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Multiple sclerosis (Nervous system disorders) | 2 | 3 | 5 | 0 | 0 | 2
Multiple sclerosis relapse (Nervous system disorders) | 0 | 1 | 5 | 0 | 0 | 2
Muscle spasticity (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Myelitis transverse (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nystagmus (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Optic neuritis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Paraparesis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Peroneal nerve palsy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Primary progressive multiple sclerosis (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Progressive multiple sclerosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Quadriparesis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Status epilepticus (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0
Trigeminal neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Uhthoff's phenomenon (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0
VIIth nerve paralysis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Adjustment disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Aggression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 2 | 0 | 1 | 0
Depressive symptom (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Mania (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Mood swings (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Panic attack (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 2 | 0 | 0 | 0
Bladder neck sclerosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nephrogenic diabetes insipidus (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 2 | 1 | 0 | 1 | 0
Neurogenic bladder (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Urethral obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 0 | 0
Adenomyosis (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Adnexal torsion (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 2 | 0 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Jessner's lymphocytic infiltration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Lentigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Activities of daily living impaired (Social circumstances) | 0 | 0 | 0 | 0 | 0 | 1
Poor personal hygiene (Social circumstances) | 1 | 0 | 0 | 0 | 0 | 0
Aneurysm (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Arterial spasm (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0
Femoral artery occlusion (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Peripheral venous disease (Vascular disorders) | 0 | 4 | 2 | 0 | 0 | 0
Raynaud's phenomenon (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Core: FTY720 1.25 mg (N=147) | Core: FTY720 0.5 mg (N=336) | Core: Placebo (N=487) | Extension: FTY1.25-0.5 (N=74) | Extension: FTY0.5-0.5 (N=196) | Extension: Placebo-FTY0.5 (N=301)
Lymphopenia (Blood and lymphatic system disorders) | 13 | 19 | 0 | 4 | 7 | 11
Abdominal pain upper (Gastrointestinal disorders) | 3 | 17 | 12 | 0 | 1 | 2
Constipation (Gastrointestinal disorders) | 10 | 27 | 35 | 0 | 2 | 6
Diarrhoea (Gastrointestinal disorders) | 13 | 15 | 18 | 1 | 3 | 1
Nausea (Gastrointestinal disorders) | 14 | 21 | 19 | 2 | 1 | 4
Fatigue (General disorders) | 16 | 24 | 43 | 0 | 1 | 9
Gait disturbance (General disorders) | 10 | 15 | 24 | 0 | 1 | 0
Pyrexia (General disorders) | 8 | 18 | 20 | 3 | 0 | 4
Bronchitis (Infections and infestations) | 10 | 16 | 21 | 3 | 2 | 1
Cystitis (Infections and infestations) | 10 | 9 | 17 | 0 | 0 | 2
Gastroenteritis (Infections and infestations) | 10 | 12 | 22 | 0 | 3 | 3
Influenza (Infections and infestations) | 14 | 26 | 43 | 3 | 4 | 9
Nasopharyngitis (Infections and infestations) | 40 | 78 | 135 | 9 | 10 | 23
Upper respiratory tract infection (Infections and infestations) | 21 | 37 | 57 | 6 | 6 | 14
Urinary tract infection (Infections and infestations) | 21 | 47 | 75 | 4 | 11 | 25
Fall (Injury, poisoning and procedural complications) | 31 | 47 | 91 | 6 | 5 | 13
Alanine aminotransferase increased (Investigations) | 17 | 39 | 7 | 0 | 1 | 6
Blood cholesterol increased (Investigations) | 8 | 15 | 16 | 0 | 1 | 3
Gamma-glutamyltransferase increased (Investigations) | 19 | 31 | 3 | 0 | 3 | 5
Hypercholesterolaemia (Metabolism and nutrition disorders) | 10 | 13 | 19 | 4 | 4 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 30 | 48 | 3 | 3 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 36 | 75 | 5 | 5 | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 21 | 35 | 3 | 3 | 3
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 21 | 16 | 31 | 4 | 3 | 9
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 12 | 14 | 1 | 3 | 4
Dizziness (Nervous system disorders) | 10 | 19 | 29 | 2 | 0 | 2
Headache (Nervous system disorders) | 28 | 56 | 77 | 3 | 3 | 13
Depression (Psychiatric disorders) | 11 | 15 | 37 | 2 | 2 | 4
Insomnia (Psychiatric disorders) | 8 | 12 | 29 | 1 | 4 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 28 | 34 | 2 | 1 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 14 | 16 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 8 | 15 | 19 | 2 | 1 | 6
Hypertension (Vascular disorders) | 23 | 43 | 28 | 2 | 5 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety